CLINICAL TRIAL: NCT04150744
Title: Radiofrequency Ablation Plus Carrizumab vs Carrizumab Alone for Moderate or Advanced Hepatocellular Carcinoma: A Real World Study
Brief Title: RFA Plus Carrizumab vs Carrizumab Alone for HCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1102320191018
Record Dates: First submitted 2019-10-28; First posted 2019-11-05 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2019-10

CONDITIONS: Tumor Immunity; Immunosuppression; Radiofrequency Ablation
Keywords: RFA; immunosuppressant; hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RFA plus carrizumab (Experimental)
  Interventions: Combination Product: radiofrequency ablation
- carrizumab (Placebo Comparator)
  Interventions: Combination Product: radiofrequency ablation

INTERVENTIONS:
Combination Product: radiofrequency ablation — take advantage of RFA to destroy hepatocellular carcinoma by high temperature

SUMMARY:
The study aims to find whether patients with advanced HCC can get more benefits from RFA +PD-1 immunosuppressant (carrizumab) compared with carrizumab alone, considering with the result of PFS.

DETAILED DESCRIPTION:
The study aims to find whether patients with advanced HCC can get more benefits from RFA +PD-1 immunosuppressant (carrizumab) compared with carrizumab alone, considering with the result of PFS. 120 patients were enrolled into two groups respectively, the experimental group and reference group.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18-75 years
2. Diagnosis as hepatocellular carcinoma from histology and cytology
3. BCLC B-C degree
4. Score of ECOG PS: 0-2
5. Child-Pugh Score: A or B
6. Not suitable for resection or liver transplantation
7. Have not received systemic therapy
8. Have at least one evaluable target mass from CT or MRI according to mRECIST
9. The estimated survival time ≥ 12 weeks
10. Patients with HBV infection having HBV-DNA <500IU/mL and standard anti-virus treatment. Patients with HCV infection must receive standard anti-virus treatment.
11. The function of main organs normal
12. Sign informed consent

Exclusion Criteria:

1. Have cholangiocarcinoma, mixed type of hepatocarcinoma and fibrolamellar hepatocellular carcinoma. Have incurable malignant tumor in five years.
2. Have local ablation, TACE or radiotherapy in 3 months before enrolled.
3. Prepared to or have received organic or bone marrow transplantation.
4. Uncontrollable ascites, hepatic encephalopathy or esophageal and gastric varices.
5. Have hypertension and can't lower down to the normal level using blood pressure medication.
6. Have type II myocardial ischemia or myocardial infarction, uncontrollable arrhythmia.
7. Have diseases to influent the effect of oral drugs, for example, unable to swallow, chronic diarrhea and intestinal obstruction.
8. Have gastrointestinal bleeding in 6 months
9. Have abdominal fistula, gastrointestinal perforation or abdominal abscess
10. Patients with lung fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug related pneumonia or severe dysfunction of lung.
11. Routine urine test showed urinary protein ≥++ or the 24 hours amount of urinary protein ≥1.0 g
12. Patients have autoimmune disease
13. Patients need corticosteroid or other immunosuppressant therapy
14. Patients have anti-tumor vaccine and other immunostimulate anti-tumor drugs in 3 months
15. Allergy to monocloning antibody
16. Pregnant or breastfeeding female Other patients not suitable to be enrolled in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | through study completion, an average of 4 years
  Time from patients received treatment fist time to disease progress or death

SECONDARY OUTCOMES:
Objective response rate | through study completion, an average of 4 years
  The ratio of patients with regressive disease ,including complete response and partial response
Disease control rate | through study completion, an average of 4 years
  The ratio of patients with regressive or stable disease, including complete response, partial response and stable disease.
Overall survival | through study completion, an average of 4 years
  Time from the random assignment to death (the last follow-up time for patients lost to follow-up, the end of study for patients still alive
Duration of response | through study completion, an average of 4 years
  Time from the first time of complete regression or partial regression to progressive disease or death

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Tang, Dr., Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- the Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No